CLINICAL TRIAL: NCT01314976
Title: Metronidazole for the Treatment of Dientamoebiasis in Children in Denmark - A Randomized, Placebo-controlled, Double-blinded Clinical Trial
Brief Title: Treatment Study of Metronidazole to Treat Dientamoebiasis in Children
Acronym: DFPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Statens Serum Institut (Other)
Responsible Party: Principal Investigator, Dennis Roser, MD, PhD fellow, Statens Serum Institut
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DSR-01; 2010-024657-36 (EudraCT Number)
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Dientamoebiasis
Keywords: Children; parasite; intestinal; treatment; RCT
MeSH Terms: conditions — Dientamoebiasis | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metronidazole (Experimental): Active treatment.
  Interventions: Drug: Metronidazole
- Placebo (Placebo Comparator): Passive treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metronidazole — Metronidazole, oral suspension, 40mg/ml.
  1 treatment period of 40mg/kg/day for 10 days, 3 daily dosages. Administered by parents.
  Other Names: Flagyl® (Metronidazole), oral suspension. Sanofi-aventis; ATC-code: P01AB01
  Arms: Metronidazole
Drug: Placebo — Placebo.
  1 treatment period of 1ml/kg/day for 10 days, 3 daily dosages. Administered by parents.
  Placebo formulation is identical to Flagyl® (Metronidazole), oral suspension from Sanofi-Aventis.
  Arms: Placebo

SUMMARY:
Introduction: Dientamoeba fragilis (DF) is a commonly occurring intestinal protozoan that is considered a possible cause of infectious gastrointestinal disease in adults and children. DF has a particular high prevalence in children, and it is suspected that children present more symptoms in infection than adults. However, evidence of causality is lacking, treatment regimens are largely untested in controlled trials, and the most commonly used antibiotic against DF in Denmark, metronidazole, has never been tested against placebo.

Main objective: To determine the clinical effect of metronidazole in DF-infected children with gastrointestinal complaints, where no other aetiology is known and no other gastrointestinal pathogens could be shown.

ELIGIBILITY:
Inclusion Criteria:

* Patients with samples investigated at Statens Serum Institut.
* Faecal sample (index) positive for Dientamoeba fragilis (DF) by realtime PCR, within < 7 days.
* No faecal samples positive for DF within the period: 3 months prior to and up to index-sample.
* Telephone interview to parents no later then 14 days after result from index-sample.
* Age 3-12 years old.
* Place of residence: Island of Zealand, incl. capital region.
* Symptoms consistent with gastrointestinal infection of DF: Either 1) ≥ 2 episodes of diarrhea per week or 2) ≥ 2 episodes of stomach ache per week or 3) ≥ 2 of the following symptoms: Anorexia, Failure to thrive, Anal itching, excessive flatulence, other change in bowel movements.

Exclusion Criteria:

* Expected non-compliance.
* Objection to subject participation from referring physician.
* Underlying illness or comorbidity, incl. known gastrointestinal illness (both infectious and non-infectious), but excluding constipation.
* Known liver disease or intolerance/allergy to metronidazole.
* Positive screening for other intestinal pathogens, which may explain subject symptoms.
* Treatment with metronidazole outside of study within study period.
* Weight > 50 kg

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Overall gastrointestinal symptoms, day 14 | 14 days after end of treatment period
  All participants receive 10 days of treatment with study drug (placebo or active). Primary outcome measure is registered on day 14 after end of treatment, using a questionnaire for the parents of the study participant.
  Measuring will be done using a VAS-score scale, addressing overall level of gastrointestinal symptoms in the previous 14 days. Results will be noted as a value from 0 to 10.

SECONDARY OUTCOMES:
Realtime PCR for D. fragilis, day 14 | Sample collection 14 days after end of treatment period
  Secondary outcome measure will be registered using a specific realtime PCR for D. fragilis, performed on faecal samples collected from study-participant.
  Results will be noted as either positive or negative.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Röser, MD, Principal Investigator — Statens Serum Institut; Dennis Röser, MD, Study Director — Statens Serum Institut
Locations (1):
- Statens Serum Institut, Copenhagen, Denmark

REFERENCES:
- [Derived] Roser D, Simonsen J, Stensvold CR, Olsen KE, Bytzer P, Nielsen HV, Molbak K. Metronidazole therapy for treating dientamoebiasis in children is not associated with better clinical outcomes: a randomized, double-blinded and placebo-controlled clinical trial. Clin Infect Dis. 2014 Jun;58(12):1692-9. doi: 10.1093/cid/ciu188. Epub 2014 Mar 18. PMID 24647023